CLINICAL TRIAL: NCT04520906
Title: Prospective, Multicenter, Single-group Target Study to Evaluate the Safety and Efficacy of Microwave Ablation Therapy in Patients With Primary Liver Cancer
Brief Title: To Evaluate the Safety and Efficacy of Microwave Ablation Therapy in Patients With Primary Liver Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Obtaining medical device market approval through the predicate device comparison route.
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MWA1.0
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, single-group target value
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental): Subjects will be treated with microwave ablation.
  Interventions: Device: microwave ablation

INTERVENTIONS:
Device: microwave ablation — ultrasound-guided microwave ablation is performed to treat hepatocellular carcinoma patients

SUMMARY:
Through the implementation of prospective, multi-center, single-group target value research to verify the safety and effectiveness of the microwave ablation treatment system for the ablation treatment of primary liver cancer.

DETAILED DESCRIPTION:
The safety and effectiveness of the microwave ablation treatment system produced by Suzhou Hengrui Hongyuan Medical Technology Co., Ltd. for the ablation treatment of primary liver cancer is verified through the implementation of prospective, multi-center, single-group target value research. According to the requirements of the trial, 139 patients who were diagnosed with primary liver cancer before surgery and met the inclusion criteria without any exclusion criteria were selected for treatment of their liver cancer with a microwave ablation treatment system, 1 month, 3 months and 6 months after surgery Carry out clinical and imaging follow-up to evaluate the safety of the operation and the effect of tumor ablation.

ELIGIBILITY:
Inclusion Criteria:

* Pathological and/or clinical diagnosis confirmed as primary liver cancer (hepatocellular carcinoma).
* Single tumor with maximum diameter ≤ 5cm ; or tumors number ≤ 3 with maximum diameter ≤ 3cm.
* No invasion of blood vessels, gallbladder, adjacent organs and distant metastasis.
* Child-Pugh class A or B classification, or meet the standard after treatment.
* Able to understand the content of clinical trials, voluntarily participate in the trial and sign informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding, or preparing to become pregnant during the trial.
* Participating in clinical trials of other devices or drugs.
* Uncorrectable coagulation dysfunction (after corrective treatment, the PT exceeds the normal control value by more than 3s).
* PLT <50x109/L.
* Intractable massive ascites.
* Cachexia.
* MRI examination is contraindicated or the investigator judges it is not suitable for MRI examination.
* Patients with bleeding from esophageal (fundus of stomach) varicose veins 1 month before surgery.
* Patients with impaired consciousness or unable to cooperate with treatment.
* The investigator judged that it is not suitable to participate in clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Complete tumor ablation rate | 1 month after surgery
  the percentage of complete ablation subjects for all subjects undergoing ablation surgery.
  Complete ablation: Follow up by MRI scan 1 month after surgery, the area where the tumor is located is in the low-density arterial phase without enhancement; if the tumor is followed up by MRI scan 1 month after surgery, there is enhancement in the local arterial phase within the tumor lesion, which suggests that the tumor remains. The tumor could be treated by re-ablation; if there is still residual tumor in MRI scan 1 month after the second ablation, it is judged as incomplete ablation.

SECONDARY OUTCOMES:
First complete tumor ablation rate | 1 month after surgery
  the percentage of subjects who did not undergo the second one month after the operation accounted for all the ablation trials.
Complete ablation rate of lesions | 1 month after surgery
  the percentage of lesions that are completely ablated to all lesions undergoing ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, Doctor, Principal Investigator — Zhongda Hospital
Locations (13):
- China (13):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - Ruijin Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Central Hospital of Lishui City, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No